CLINICAL TRIAL: NCT00330941
Title: Intravenous Lidocaine Infusion Improves Outcome After Laparoscopic Colectomy
Brief Title: Intravenous Lidocaine and Acute Rehabilitation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: University of Liege (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Joris, Lidocaine Outcomes
Record Dates: First submitted 2006-05-25; First posted 2006-05-29 (Estimated); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Pain, Postoperative; Opioid Consumption, Postoperative; Postoperative Fatigue
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine

INTERVENTIONS:
Drug: lidocaine

SUMMARY:
Background: Intravenous infusion of lidocaine may decrease postoperative pain and speed return of bowel function. The investigators therefore tested the hypothesis that including perioperative lidocaine infusion improves recovery from laparoscopic colectomy and shortens the duration of hospitalization.

Methods: Forty patients scheduled for laparoscopic colectomy were randomly allocated to receive intravenous lidocaine (bolus injection of 1.5 mg.kg-1 lidocaine at induction of anesthesia, then a continuous infusion of 2 mg.kg-1.h-1 intraoperatively and 1.33 mg.kg-1.h-1 for 24 h postoperatively) or an equal volume of saline. All patients received similar intensive postoperative rehabilitation. Postoperative pain scores, opioid consumption, and fatigue scores were measured. Times to first flatus, defecation, and hospital discharge were recorded. Postoperative endocrine (cortisol and catecholamines) and metabolic (leucocytes, C-reactive protein, and glucose) responses were measured for 48 h. Data (median [25%-75% interquartile range] Saline vs Lidocaine groups) were analyzed using Mann-Whitney tests. P<0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* non-malignant disease

Exclusion Criteria:

* greater than 70 years
* history of gastro-duodenal peptic ulcer or renal failure (contraindications to the use of nonsteroidal anti-inflammatory drug)
* hepatic insufficiency
* psychiatric disorder
* steroid treatment
* chronic treatment with opioid

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2003-01; Study Completion 2004-12

PRIMARY OUTCOMES:
Sevoflurane consumption
Pain scores
abdominal comfort
fatigue scores

SECONDARY OUTCOMES:
bowel function
hospital stay
endocrine and metabolic responses

CONTACTS AND LOCATIONS:
Overall Officials: Jean Joris, MD, PhD, Study Director — Department of Anesthesia and Intensive Care Medicine, CHU de Liège, University of Liège, Belgium
Locations (1):
- CHU de Liège, University of Liège, Liège, Belgium